CLINICAL TRIAL: NCT00814905
Title: Treatment of Chorioamnionitis After Delivery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI retired
Sponsor: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PO8-098
Record Dates: First submitted 2008-12-23; First posted 2008-12-25 (Estimated); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Chorioamnionitis
Keywords: chorioamnionitis; antibiotics; cesarean; vaginal delivery
MeSH Terms: conditions — Chorioamnionitis | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- vaginal delivery 1 (Placebo Comparator): no further antibiotics after delivery (the patient will receive a saline infusion instead of antibiotics)
  Interventions: Drug: saline
- vaginal delivery antibotics2 (Active Comparator): one additional dose of antibiotics (ampicillin 2 grams IV, gentamicin 1.5 mg/kg IV) following vaginal delivery
  Interventions: Drug: ampicillin gentamicin
- cesarean delivery one dose3 (Other): one dose of ampicillin 2 grams IV, gentamicin 1.5 mg/kg IV, clindamycin 900 mg IV and then saline infusions instead of antibiotics until they are afebrile for 24 hours ( they will receive saline infusions instead of antibiotics)
  Interventions: Drug: Ampicillin gentamicin clindamycin
- cesarean multiple antibiotics 4 (Other): ampicillin 2 g IV every 6 hours, gentamicin 1.5mg/kg every 8 hours, and clindamycin 900 mg IV every 8 hours until the patient has been afebrile for 24 hours
  Interventions: Drug: ampicillin gentamicin clindamycin

INTERVENTIONS:
Drug: saline — A saline infusion after delivery (one dose)
  Arms: vaginal delivery 1
Drug: ampicillin gentamicin — one additional dose of antibiotics (ampicillin 2 grams IV, gentamicin 1.5 mg/kg IV) following their vaginal delivery
  Arms: vaginal delivery antibotics2
Drug: Ampicillin gentamicin clindamycin — one dose of ampicillin 2 grams IV, gentamicin 1.5 mg/kg IV, clindamycin 900 mg IV and then saline infusions instead of antibiotics until they are afebrile for 24 hours ( they will receive saline infusions instead of antibiotics)
  Arms: cesarean delivery one dose3
Drug: ampicillin gentamicin clindamycin — ampicillin 2 g IV every 6 hours, gentamicin 1.5mg/kg every 8 hours, and clindamycin 900 mg IV every 8 hours until the patient has been afebrile for 24 hours
  Arms: cesarean multiple antibiotics 4

SUMMARY:
Chorioamnionitis occurs in 1% to 5% of term pregnancies and may complicate up to 25% of cases of preterm labor. The traditional regimen used to treat intra-amniotic infection is intravenous ampicillin 2g every 6 hours and intravenous gentamicin 1.5 mg/kg every 8 hrs until delivery . In the past the recommendation has been that the antibiotics be continued postpartum until 24-48 hours afebrile. More recent studies have looked at using a one time dose of antibiotics after delivery vs treating until 24-48 hours afebrile. There have been no studies comparing treatment of chorioamnionitis with antibiotics vs no treatment with antibiotics postpartum. The aim of this study is to compare no treatment vs treatment with one dose after a vaginal delivery and one dose of antibiotics vs a full course until 24 hours afebrile after a cesarean delivery complicated by chorioamnionitis. The hypothesis is that there will be no difference in outcome between the two groups in each arm. This is a randomized study. Once the patient delivers she will be randomized to one of two groups in each arm. First arm (vaginal delivery) A: no treatment, B: treatment with a one time dose of ampicillin/gentamicin; Second arm (c/s) A: one dose of ampicillin/gentamicin/clindamycin, B: treatment with ampicillin/gentamicin and clindamycin until 24 hours afebrile. The goal of the study is to determine the optimal postpartum management of chorioamnionitis.

DETAILED DESCRIPTION:
Chorioamnionitis refers to infection of the amniotic fluid, membranes, placenta and/or uterus. Clinical chorioamnionitis is defined by a temperature of 380 C or more and one or more of the following findings: maternal heart rate > 100 BPM, baseline fetal heart rate > 160 BPM, uterine tenderness, or foul smelling amniotic fluid. It complicates 0.5 to 10.5 percent of deliveries and accounts for 10 to 40 percent of cases of maternal febrile morbidity in the peripartum period and 50 percent of preterm deliveries before 30 weeks of gestation. Chorioamnionitis is also associated with 20 to 40 percent of cases of early neonatal sepsis and pneumonia. (Hagberg et al). The most extensively tested antibiotic regimen is ampicillin 2 g IV every 6 hours and gentamicin 1.5mg/kg every 8 hours. After delivery clindamycin 900 mg IV q 8 hours can be used for further coverage in those women delivering by cesarean section. The treatment is usually continued until the patient is asymptomatic for 24 - 48 hours although that treatment is primarily based on expert opinion. (Edwards et al). Potential benefits of not needing to treat with antibiotics after a delivery complicated by intramniotic infection is shortened hospital stay and reduced cost. No studies up until now have compared treatment verses no treatment head to head for vaginal delivery and one postpartum dose vs. continued treatment for 24 hours in the women undergoing a cesarean delivery. Unfortunately the Duff study combined patients analyzing both vaginal deliveries and cesarean deliveries together. They were both treated with either the single dose of antibiotics or continual treatment with antibiotics until afebrile and asymptomatic for 24 hours. He found no statistical significant difference in treatment failure in the one dose vs. multiple dose groups. This finding was the primary outcome of the study.Our study will be a double blind placebo controlled randomized study. There will be two arms: vaginal delivery and cesarean delivery. The first arm consists of patients who have had a vaginal delivery complicated by chorioamnionitis. They will be randomized into one of two groups: 1) no further antibiotics after delivery ( they will receive a saline infusion instead of antibiotics but this will be labeled in the pharmacy and neither the patient nor the physician will know whether the patient is receiving antibiotics or saline) or 2) one additional dose of antibiotics (ampicillin 2 grams IV, gentamicin 1.5 mg/kg IV) following their vaginal delivery. The second arm of this study consists of patients who have had a cesarean delivery complicated by chorioamnionitis. They will also be randomized into one of two groups: 1) one dose of ampicillin 2 grams IV, gentamicin 1.5 mg/kg IV, clindamycin 900 mg IV and then saline infusions instead of antibiotics until they are afebrile for 24 hours ( they will receive saline infusions instead of antibiotics but this will be labeled in the pharmacy and neither the patient or the physician will know whether the patient is receiving antibiotics or saline) or 2) ampicillin 2 g IV every 6 hours, gentamicin 1.5mg/kg every 8 hours, and clindamycin 900 mg IV every 8 hours until the patient has been afebrile for 24 hours. For the patients in both arms of the study the primary outcome will be treatment failure defined as either a single temperature of 39 C or two or more temperatures of 38.4 C or more at least 4 hours apart after delivery in the vaginal group or after the first antibiotic dose in the cesarean group. All treatment failures will be treated with ampicillin 2 grams IV every 6 hours, gentamicin 1.5 mg/kg every 8 hours and clindamycin 900 mg every 8 hours until the patient has been afebrile and asymptomatic for 24 hours. Timing of temperature spikes or other symptoms associated with uterine infection will be noted as well as number of doses of antibiotics and infection related complications such as wound infection, pelvic abscess and septic pelvic thrombophlebitis. Patients will be recruited from the Labor and Delivery unit here at Naval Medical Center Portsmouth. All patients that develop chorioamnionitis will be offered participation in the study. All women greater than 18 years old will be eligible to participate. Patients will be consented by the residents and staff working on labor and delivery. Exclusion criteria will include those who do not wish to participate, patients who are allergic to the study antibiotics, women who are immunocompromised or women receiving antibiotics for other reasons such as prophylaxis for bacterial endocarditis.

ELIGIBILITY:
Inclusion Criteria:.

* All patients that develop chorioamnionitis and who are over 18 years of age will be offered participation in the study.

Exclusion Criteria:

* Women who do not wish to participate, patients who are allergic to the study antibiotics
* Women who are immunocompromised or women receiving antibiotics for other reasons such as prophylaxis for bacterial endocarditis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11-18 (Actual); Primary Completion 2012-01 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
To determine the courses of antibiotics needed after vaginal delivery and after cesareans in pregnancies complicated by chorioamnionitis. | Postpartum 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Everett F Magann, MD, Principal Investigator — Naval Officer, Naval Medical Center - Portsmouth
Locations (1):
- Naval Medical Center - Portsmouth, Portsmouth, Virginia, United States